CLINICAL TRIAL: NCT00473694
Title: A Multicenter, Randomized, Parallel Group Comparative, Active-Controlled, Safety-assessor Blinded. Phase IIIa, Pivotal Trial in Adult Subjects Comparing Org 25969 With Neostigmine as Reversal Agent of a Neuromuscular Block Induced by Maintenance Dosing of Rocuronium or Vecuronium at 1-2 PTCs
Brief Title: Comparison of Sugammadex (MK-8616/Org 25969) With Neostigmine Administered at 1-2 Post-tetanic Counts (PTCs) After Administration of Rocuronium or Vecuronium (19.4.302/P05945/MK-8616-025)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P05945; 19.4.302 (Other: Organon Protocol Number); P05945 (Other: Schering-Plough Protocol Number); MK-8616-025 (Other: Merck Protocol Number)
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex; Neostigmine; Vecuronium Bromide; Rocuronium; Glycopyrrolate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- rocuronium+sugammadex (Experimental): Participants received a single bolus dose of 0.60 mg/kg rocuronium prior to intubation. The neuromuscular block was maintained with 0.15 mg/kg rocuronium if needed. At 1-2 post-tetanic counts (PTC) and after the last dose of rocuronium, a single bolus dose of 4.0 mg/kg sugammadex was administered.
  Interventions: Drug: sugammadex; Drug: rocuronium
- rocuronium+neostigmine (Active Comparator): Participants received a single bolus dose of 0.60 mg/kg rocuronium prior to intubation. The neuromuscular block was maintained with 0.15 mg/kg rocuronium if needed. At 1-2 PTC and after the last dose of rocuronium, a single bolus dose of 70.0 μg/kg neostigmine (up to a maximum dose of 5 mg) was administered in combination with 14.0 μg/kg glycopyrrolate.
  Interventions: Drug: neostigmine; Drug: rocuronium; Drug: glycopyrrolate
- vecuronium+sugammadex (Experimental): Participants received a single bolus dose of 0.1 mg/kg vecuronium prior to intubation. The neuromuscular block was maintained with 0.015 mg/kg vecuronium if needed. At 1-2 PTC and after the last dose of vecuronium, a single bolus dose of 4.0 mg/kg sugammadex was administered.
  Interventions: Drug: sugammadex; Drug: vecuronium
- vecuronium+neostigmine (Active Comparator): Participants received a single bolus dose of 0.1 mg/kg vecuronium prior to intubation. The neuromuscular block was maintained with 0.015 mg/kg vecuronium if needed. At 1-2 PTC and after the last dose of vecuronium, a single bolus dose of 70.0 μg/kg neostigmine (up to a maximum dose of 5 mg) was administered in combination with 14.0 μg/kg glycopyrrolate.
  Interventions: Drug: neostigmine; Drug: vecuronium; Drug: glycopyrrolate

INTERVENTIONS:
Drug: sugammadex — Administered as an intravenous (IV) infusion
  Other Names: Org 25969; MK-8616; BRIDION®
  Arms: rocuronium+sugammadex; vecuronium+sugammadex
Drug: neostigmine — Administered as an IV infusion
  Other Names: PROSTIGMIN®
  Arms: rocuronium+neostigmine; vecuronium+neostigmine
Drug: vecuronium — Administered as an IV infusion
  Other Names: NORCURON®
  Arms: vecuronium+neostigmine; vecuronium+sugammadex
Drug: rocuronium — Administered as an IV infusion
  Other Names: ZEMURON®
  Arms: rocuronium+neostigmine; rocuronium+sugammadex
Drug: glycopyrrolate — Administered as an IV infusion
  Other Names: ROBINUL®
  Arms: rocuronium+neostigmine; vecuronium+neostigmine

SUMMARY:
The purpose of the trial is to demonstrate a faster recovery from neuromuscular block (NMB) induced with rocuronium or vecuronium after reversal by 4.0 mg/kg of Org 25969 compared with reversal by 70 μg/kg of neostigmine in combination with 14 μg/kg glycopyrrolate.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class 1 to 4
* 18 years or older
* Scheduled to undergo an elective surgical procedure under general anesthesia requiring the use of rocuronium or vecuronium for endotracheal intubation and maintenance of neuromuscular block
* Scheduled for surgery in supine position
* Given written informed consent

Exclusion Criteria:

* Participants in whom a difficult intubation is expected due to anatomical malformations
* Known or suspected to have neuromuscular disorders impairing neuromuscular blockade and/or significant renal dysfunction
* Known or suspected to have a (family) history of malignant hyperthermia
* Known or suspected to have an allergy to narcotics, muscle relaxants, or other medications used during surgery
* Receiving medication known to interfere with neuromuscular blocking agents such as anticonvulsants, antibiotics, and magnesium (Mg2+)
* Participants in whom the use of neostigmine and/or glycopyrrolate may be contraindicated
* Female participants who are pregnant or breast-feeding
* Females participants of childbearing potential not using an acceptable method of birth control [condom or diaphragm with spermicide, vasectomized partner (> 6 months), IUD, abstinence]
* Participants who had already participated in an Org 25969 trial
* Participants who had participated in another clinical trial, not pre-approved by Organon, within 30 days of entering into Protocol 19.4.302

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2005-11-28 (Actual); Primary Completion 2006-11-06 (Actual); Study Completion 2007-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Lemmens HJ, El-Orbany MI, Berry J, Morte JB Jr, Martin G. Reversal of profound vecuronium-induced neuromuscular block under sevoflurane anesthesia: sugammadex versus neostigmine. BMC Anesthesiol. 2010 Sep 1;10:15. doi: 10.1186/1471-2253-10-15. PMID 20809967
- [Result] Jones RK, Caldwell JE, Brull SJ, Soto RG. Reversal of profound rocuronium-induced blockade with sugammadex: a randomized comparison with neostigmine. Anesthesiology. 2008 Nov;109(5):816-24. doi: 10.1097/ALN.0b013e31818a3fee. PMID 18946293
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 8 trial sites in the United States. A total of 182 participants were randomized with 157 participants treated.
Groups:
- Rocuronium+Neostigmine: Participants received a single bolus dose of 0.60 mg/kg rocuronium prior to intubation. The neuromuscular block was maintained with 0.15 mg/kg rocuronium if needed. At 1-2 PTC and after the last dose of rocuronium, a single bolus dose of 70.0 μg/kg neostigmine (up to a maximum dose of 5 mg) was administered in combination with 14.0 μg/kg glycopyrrolate .
- Vecuronium+Neostigmine: Participants received a single bolus dose of 0.1 mg/kg vecuronium prior to intubation. The neuromuscular block was maintained with 0.015 mg/kg vecuronium if needed. At 1-2 PTC and after the last dose of vecuronium, a single bolus dose of 70.0 μg/kg neostigmine (up to a maximum dose of 5 mg) was administered in combination with 14.0 μg/kg glycopyrrolate .
Period: Overall Study
Arm/Group | Rocuronium+Sugammadex | Rocuronium+Neostigmine | Vecuronium+Sugammadex | Vecuronium+Neostigmine
Started | 48 | 41 (Includes 1 participant randomized to vecuronium+sugammadex but treated with rocuronium+neostigmine) | 51 | 42
Treated | 37 (Number of participants treated was based on actual treatment received.) | 38 (Number of participants treated was based on actual treatment received.) | 46 (Number of participants treated was based on actual treatment received.) | 36 (Number of participants treated was based on actual treatment received.)
Completed | 37 (Number of participants completed was based on actual treatment received.) | 37 (Number of participants completed was based on actual treatment received.) | 46 (Number of participants completed was based on actual treatment received.) | 35 (Number of participants completed was based on actual treatment received.)
Not Completed | 11 | 4 | 5 | 7
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Participants did not receive treatment | 11 | 3 | 5 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population was all randomized participants.
Groups:
- Rocuronium+Sugammadex: Participants received a single bolus dose of 0.60 mg/kg rocuronium prior to intubation. The neuromuscular block was maintained with 0.15 mg/kg rocuronium if needed. At 1-2 PTC and after the last dose of rocuronium, a single bolus dose of 4.0 mg/kg sugammadex was administered.
- Total: Total of all reporting groups
Arm/Group | Rocuronium+Sugammadex | Rocuronium+Neostigmine | Vecuronium+Sugammadex | Vecuronium+Neostigmine | Total
Number analyzed (Participants) | 48 | 40 | 52 | 42 | 182
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The analysis population was all randomized participants.
  Years | 53.6 (14.0) | 54.0 (10.8) | 49.9 (13.6) | 55.2 (13.3) | 53.0 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The analysis population was all randomized participants.
  Participants
    Female | 26 | 20 | 33 | 21 | 100
    Male | 22 | 20 | 19 | 21 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The analysis population was all randomized participants.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 3 | 1 | 3 | 7
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 3 | 1 | 7 | 2 | 13
    White | 43 | 36 | 43 | 37 | 159
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 2 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Administration of Sugammadex or Neostigmine to Recovery of the T4/T1 Ratio to 0.9 After Neuromuscular Block (NMB) Induced by Rocuronium
Description: Mean time from start of sugammadex or neostigmine administration to recovery of T4/T1 ratio to 0.9 was assessed by applying repetitive train of four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. Nerve stimulation continued until the ratio of the magnitude of the fourth twitch (T4) to first twitch (T1) reached at least 0.9. The greater the T4/T1 ratio represented the greater the recovery from NMB; with a value of 0.0 representing no recovery and 1.0 representing full recovery. Reduced recovery time of the T4/T1 ratio to 0.9 indicated faster recovery from NMB. Mean time was collected in minutes and seconds but converted to and presented in minutes only. The analysis included a procedure for the imputation of missing recovery times.
Time Frame: Up to approximately 3 hours after administration of study drug
Population: The analysis population was the Intent-to-Treat population that included all participants who received study drug and had at least one post-baseline efficacy assessment and were analyzed in the group to which they were randomized (initial treatment assignment and not by the actual treatment received).
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium+Sugammadex | Rocuronium+Neostigmine
Number analyzed (Participants) | 37 | 37
Minutes | 3.28 (2.40) | 55.50 (27.10)
Statistical Analysis 1: Comparison: Rocuronium+Sugammadex vs Rocuronium+Neostigmine; Test type: Superiority; p < 0.0001, ANOVA — A two-way ANOVA model was used with the logarithm of the recovery time taken as the response variable, and trial site and treatment group were the factors of the model; Estimated Treatment Effect = 17.29, 95% CI 2-sided [13.95 to 21.42] — The value for estimated treatment effect represents how many times faster the mean time to recovery of the T4/T1 ratio to 0.9 was for participants receiving sugammadex after NMB compared to participants receiving neostigmine after NMB

2. Primary Outcome: Time From Start of Administration of Sugammadex or Neostigmine to Recovery of the T4/T1 Ratio to 0.9 After Neuromuscular Block (NMB) Induced by Vecuronium
Description: as for outcome 1
Time Frame: Up to approximately 6 hours after administration of study drug
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Vecuronium+Sugammadex | Vecuronium+Neostigmine
Number analyzed (Participants) | 47 | 36
Minutes | 8.73 (14.60) | 77.80 (56.98)
Statistical Analysis 1: Comparison: Vecuronium+Sugammadex vs Vecuronium+Neostigmine; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Estimated Treatment Effect = 14.86, 95% CI 2-sided [10.18 to 21.67] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time From Start of Administration of Sugammadex or Neostigmine to Recovery of the T4/T1 Ratio to 0.7 After Neuromuscular Block (NMB) Induced by Rocuronium
Description: Mean time from start of sugammadex or neostigmine administration to recovery of T4/T1 ratio to 0.7 was assessed by applying repetitive train of four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. Nerve stimulation continued until the ratio of the magnitude of the fourth twitch (T4) to first twitch (T1) reached at least 0.7. The greater the T4/T1 ratio represented the greater the recovery from NMB; with a value of 0.0 representing no recovery and 1.0 representing full recovery. Reduced recovery time of the T4/T1 ratio to 0.7 indicated faster recovery from NMB. Mean time was collected in minutes and seconds but converted to and presented in minutes only. The analysis included a procedure for the imputation of missing recovery times.
Time Frame: Up to approximately 2 hours after administration of study drug
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium+Sugammadex | Rocuronium+Neostigmine
Number analyzed (Participants) | 37 | 37
Minutes | 2.27 (1.25) | 37.68 (21.88)
Statistical Analysis 1: Comparison: Rocuronium+Sugammadex vs Rocuronium+Neostigmine; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Estimated Treatment Effect = 15.84, 95% CI 2-sided [12.58 to 19.95] — The value for estimated treatment effect represents how many times faster the mean time to recovery of the T4/T1 ratio to 0.7 was for participants receiving sugammadex after NMB compared to participants receiving neostigmine after NMB

4. Secondary Outcome: Time From Start of Administration of Sugammadex or Neostigmine to Recovery of the T4/T1 Ratio to 0.7 After Neuromuscular Block (NMB) Induced by Vecuronium
Description: as for outcome 3
Time Frame: Up to approximately 4 hours after administration of study drug
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Vecuronium+Sugammadex | Vecuronium+Neostigmine
Number analyzed (Participants) | 47 | 36
Minutes | 4.10 (8.78) | 56.17 (36.65)
Statistical Analysis 1: Comparison: Vecuronium+Sugammadex vs Vecuronium+Neostigmine; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Estimated Treatment Effect = 18.45, 95% CI 2-sided [13.98 to 24.35] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Time From Start of Administration of Sugammadex or Neostigmine to Recovery of the T4/T1 Ratio to 0.8 After Neuromuscular Block (NMB) Induced by Rocuronium
Description: Mean time from start of sugammadex or neostigmine administration to recovery of T4/T1 ratio to 0.8 was assessed by applying repetitive train of four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. Nerve stimulation continued until the ratio of the magnitude of the fourth twitch (T4) to first twitch (T1) reached at least 0.8. The greater the T4/T1 ratio represented the greater the recovery from NMB; with a value of 0.0 representing no recovery and 1.0 representing full recovery. Reduced recovery time of the T4/T1 ratio to 0.8 indicated faster recovery from NMB. Mean time was collected in minutes and seconds but converted to and presented in minutes only. The analysis included a procedure for the imputation of missing recovery times.
Time Frame: Up to approximately 3 hours after administration of study drug
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium+Sugammadex | Rocuronium+Neostigmine
Number analyzed (Participants) | 37 | 37
Minutes | 2.65 (1.58) | 45.82 (24.95)
Statistical Analysis 1: Comparison: Rocuronium+Sugammadex vs Rocuronium+Neostigmine; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Estimated Treatment Effect = 17.04, 95% CI 2-sided [13.62 to 21.31] — The value for estimated treatment effect represents how many times faster the mean time to recovery of the T4/T1 ratio to 0.8 was for participants receiving sugammadex after NMB compared to participants receiving neostigmine after NMB

6. Secondary Outcome: Time From Start of Administration of Sugammadex or Neostigmine to Recovery of the T4/T1 Ratio to 0.8 After Neuromuscular Block (NMB) Induced by Vecuronium
Description: as for outcome 5
Time Frame: Up to approximately 5 hours after administration of study drug
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Vecuronium+Sugammadex | Vecuronium+Neostigmine
Number analyzed (Participants) | 47 | 36
Minutes | 5.55 (9.87) | 67.42 (44.85)
Statistical Analysis 1: Comparison: Vecuronium+Sugammadex vs Vecuronium+Neostigmine; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Estimated Treatment Effect = 17.70, 95% CI 2-sided [12.85 to 24.38] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Number of Participants Awake and Oriented After Anesthesia (Clinical Assessment of Level of Consciousness)
Description: The number of participants who were awake and oriented was assessed as part of an overall assessment of the clinical level of consciousness by the investigator. The clinical level of consciousness was used as a measure of recovery from NMB at 2 timepoints: prior to transfer to the recovery room after extubation and prior to discharge from the recovery room. Attempts were made to arouse participants every 15 minutes with mild prodding, mild shaking, and asking questions regarding name, location, and day of the week. The assessment ended once the participant was awake and fully orientated, 24 hours, or discharged from the hospital if discharge occurs before 24 hours; whichever occurred first. Participants were given a level of consciousness based on what type of stimulation they responded to. Participants who were not cooperative with the examination were not included in the assessment.
Time Frame: Up to 24 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium+Sugammadex | Rocuronium+Neostigmine | Vecuronium+Sugammadex | Vecuronium+Neostigmine
Number analyzed (Participants) | 37 | 37 | 47 | 36
Participants
  Prior to transfer to recovery room | 26 | 20 | 27 | 20
  Prior to discharge from recovery room | 34 | 32 | 39 | 33

8. Secondary Outcome: Number of Participants Aroused With Minimal Stimulation After Anesthesia (Clinical Assessment of Level of Consciousness)
Description: The number of participants aroused with minimal stimulation was assessed as part of an overall assessment of the clinical level of consciousness by the investigator. The clinical level of consciousness was used as a measure of recovery from NMB at 2 timepoints: prior to transfer to the recovery room after extubation and prior to discharge from the recovery room. Attempts were made to arouse participants every 15 minutes with mild prodding, mild shaking, and asking questions regarding name, location, and day of the week. The assessment ended once the participant was awake and fully orientated, 24 hours, or discharged from the hospital if discharge occurs before 24 hours; whichever occurred first. Participants were given a level of consciousness based on what type of stimulation they responded to. Participants who were not cooperative with the examination were not included in the assessment.
Time Frame: Up to 24 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium+Sugammadex | Rocuronium+Neostigmine | Vecuronium+Sugammadex | Vecuronium+Neostigmine
Number analyzed (Participants) | 37 | 37 | 47 | 36
Participants
  Prior to transfer to recovery room | 9 | 11 | 12 | 8
  Prior to discharge from recovery room | 0 | 1 | 2 | 1

9. Secondary Outcome: Number of Participants Responsive Only to Tactile Stimulation After Anesthesia (Clinical Assessment of Level of Consciousness)
Description: The number of participants responsive only to tactile stimulation was assessed as part of an overall assessment of the clinical level of consciousness by the investigator. The clinical level of consciousness was used as a measure of recovery from NMB at 2 timepoints: prior to transfer to the recovery room after extubation and prior to discharge from the recovery room. Attempts were made to arouse participants every 15 minutes with mild prodding, mild shaking, and asking questions regarding name, location, and day of the week. The assessment ended once the participant was awake and fully orientated, 24 hours, or discharged from the hospital if discharge occurs before 24 hours; whichever occurred first. Participants were given a level of consciousness based on what type of stimulation they responded to. Participants who were not cooperative with the examination were not included in the assessment.
Time Frame: Up to 24 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium+Sugammadex | Rocuronium+Neostigmine | Vecuronium+Sugammadex | Vecuronium+Neostigmine
Number analyzed (Participants) | 37 | 37 | 47 | 36
Participants
  Prior to transfer to recovery room | 2 | 3 | 7 | 7
  Prior to discharge from recovery room | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Able to Perform a 5-second Head Lift
Description: The number of participants who were able to lift their head for 5 seconds was assessed by the investigator as a measure of recovery from NMB at 2 timepoints: prior to transfer to the recovery room after extubation and prior to discharge from the recovery room. The assessment was performed every 15 minutes until the first successful 5-second head lift was achieved. Participants who were not cooperative with the examination were not included in the assessment.
Time Frame: Up to 24 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium+Sugammadex | Rocuronium+Neostigmine | Vecuronium+Sugammadex | Vecuronium+Neostigmine
Number analyzed (Participants) | 37 | 37 | 47 | 36
Participants
  Prior to transfer to recovery room | 33 | 28 | 36 | 24
  Prior to discharge from recovery room | 34 | 33 | 41 | 33

11. Secondary Outcome: Number of Participants Experiencing General Muscle Weakness
Description: The number of participants experiencing general muscle weakness was assessed by the investigator as a measure of recovery from NMB at 2 timepoints: prior to transfer to the recovery room after extubation and prior to discharge from the recovery room. The assessments were performed every 15 minutes until the absence of general muscle weakness. A standardized examination form was used to determine the presence or absence of muscle weakness in various muscle groups. Participants who were not cooperative with the examination were not included in the assessment.
Time Frame: Up to 24 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium+Sugammadex | Rocuronium+Neostigmine | Vecuronium+Sugammadex | Vecuronium+Neostigmine
Number analyzed (Participants) | 37 | 37 | 47 | 36
Participants
  Prior to transfer to recovery room | 3 | 5 | 4 | 2
  Prior to discharge from recovery room | 2 | 3 | 1 | 3

ADVERSE EVENTS:
Time Frame: Up to 7 days after administration of study drug
Description: The analysis population consisted of all randomized participants who received at least one dose of the study drug (All Subjects Treated Group).
Arm/Group | Rocuronium+Sugammadex | Rocuronium+Neostigmine | Vecuronium+Sugammadex | Vecuronium+Neostigmine
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38 | 0/46 | 0/36
Serious Adverse Events (participants affected / at risk) | 2/37 | 3/38 | 2/46 | 0/36
Other Adverse Events (participants affected / at risk) | 36/37 | 37/38 | 46/46 | 33/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium+Sugammadex (N=37) | Rocuronium+Neostigmine (N=38) | Vecuronium+Sugammadex (N=46) | Vecuronium+Neostigmine (N=36)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium+Sugammadex (N=37) | Rocuronium+Neostigmine (N=38) | Vecuronium+Sugammadex (N=46) | Vecuronium+Neostigmine (N=36)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (4) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 5 (5) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Flatulence (Gastrointestinal disorders) | 6 (6) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (16) | 19 (22) | 24 (25) | 12 (13)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Retching (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 7 (8) | 9 (9) | 4 (4)
Chest discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 5 (5) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (3) | 2 (2) | 3 (3)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Gastrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Incision site complication (Injury, poisoning and procedural complications) | 9 (9) | 8 (8) | 10 (10) | 8 (8)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Post procedural nausea (Injury, poisoning and procedural complications) | 7 (8) | 5 (5) | 5 (5) | 2 (2)
Procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 6 (6) | 2 (3) | 2 (2)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 1 (2)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 26 (36) | 29 (37) | 33 (38) | 24 (37)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 4 (4) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 5 (5) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 3 (4) | 4 (4) | 12 (13) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (5)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (5) | 4 (4) | 4 (4) | 2 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 8 (8) | 7 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (5) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications including scientific papers, presentations, or other communication concerning the clinical trial must first be submitted to the Sponsor at least six weeks ahead of estimated publication or presentation, for written consent. In order to protect proprietary interests, the Sponsor shall have the right to make consent conditional upon proper representation of the interpretation of both the Sponsor and the investigator(s) in the discussion of the data in such communications.